CLINICAL TRIAL: NCT05875688
Title: The Effect of Cementation Techniques on Retention of Full Veneer Crowns; an In-vitro Study
Brief Title: Cementation Techniques; an In-vitro Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 3363809324
Record Dates: First submitted 2023-01-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Cementation Teeth; Hyperplasia; Dental Cements; Tooth Crown Fracture
Keywords: Cementation; Cementation techniques; Crowns; Glass-ionomer cement; Retention
MeSH Terms: conditions — Hyperplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Filling the crown with cement up to margins.
  Interventions: Other: Cementation Technique A
- Group B (Experimental): Applying a cement layer on all fitting surfaces.
  Interventions: Other: Cementation Technique B
- Group C (Experimental): Applying a cement layer on all fitting surfaces except occlusal surface.
  Interventions: Other: Cementation Technique C

INTERVENTIONS:
Other: Cementation Technique A — * Use of adequate amount of cement.
  * Prevention of wastage of cement.
  * Retention of crowns for longer duration.
  Arms: Group A
Other: Cementation Technique B — * Use of Sufficient Cement Quantity.
  * Keeping cement from going to waste.
  * Increased time that crowns remain in place.
  Arms: Group B
Other: Cementation Technique C — * The utilisation of an appropriate quantity of cement.
  * The mitigation of cement waste.
  * Prolonged retention of dental crowns.
  Arms: Group C

SUMMARY:
The goal of this observational study invitro study was to compare the different cementation techniques used to lute full veneer crowns on extracted and prepared teeth using Glass Ionomer Cement type 1.

The main question[s] it aims to answer are:

The in-vitro effect cement application techniques on retention of full veneer crowns.

Which of the three different cementation techniques in-vitro provide a greater retention for a full veneer crown and will it achieve better retention using the concluded method for longer duration of cemented crown in oral cavity.

To use of adequate amount of cement to avoid wastage. The principal investigator applied the Glass ionomer cement in three different techniques on custom prepared crowns and with the help of an Universal Testing Machine debonded the crown from the prepared tooth. The results were compared amongst the three categories and the technique C, proved to be the superlative amongst the three.

DETAILED DESCRIPTION:
1. Tooth selection The procedure started by informing the oral surgery department to reserve mandibular premolar teeth that were being extracted each day, followed by taking patient consent for the purpose of research. The extracted teeth collected were kept in hydrogen peroxide for 5 minutes and then washed under tap water for any visible debris. The teeth were then stored in Formalin 10% for a period of 7-days, as per Centers for Disease Control and Prevention disinfection protocols. The teeth were then transported in Hanks Balanced Salt solution to maintain disinfection and tooth quality.
2. Preparation of tooth mounts The extracted teeth were then mounted in an acrylic block using self-cure acrylic resin (Shofu self cure acrylic resin, Japan). 0.5 mL of liquid was dispensed into a mixing cup, then 1 g of powder was added and quickly mixed using a spatula for 10 - 15 sec. Preformed plastic cylinders (Height; 55mm, Diameter; 20mm) were used, and inner walls painted with petroleum jelly for easy removal. The extracted teeth were then inserted in these cylinders filled with acrylic dough. Following manufacturer's instructions, it was ensured that the entire procedure was completed within 2 minutes after mixing was finished and at room temperature. The moulds were then left for an hour at room temperature to ensure complete chemical curing.
3. Crown preparation Following complete chemical cure the teeth were prepared using a high-speed handpiece with water irrigation with diamond bur (Head Diameter: 1.2mm, Head Length: 7.7mm, 06-125µmm). They were first reduced in occlusal anatomical planes and a chamfer finish line (approximately 0.75mm) was given all around. Total Occlusal Convergence was kept at 20◦ and 25◦ with a clinical height of 5mm. Preparation dimensions (Total Occlusal Convergence, height) of the teeth were checked using computer software (AutoCAD 2000) after taking pictures with digital single-lens reflex camera with 105mm lens at 100mm. The distance was reproduced using a standard metal scale. The tooth mounts were labelled and kept in Hank's Balanced Salt Solution to maintain tissue health. Any tooth that did not meet the preparation requirements was discarded according to the Centers for Disease Control and Prevention criteria.

   The data collection was performed by the principal investigator. Dental photograph measurements were initially performed by the supervisor. To avoid the photographic error the photographs were calibrated by measuring the prepared tooth and scaling it on the AutoCAD software. The complete photography setup was stationary during the data collection process. Then, the data between the two operators were subjected to correlation analysis, and a strong correlation value was found (0.839). Furthermore, 20% of photographs were then re- assessed after a period of 2 weeks by the same operator. The data was analyzed later by formula to confirm intra-operator reliability through correlation statistics. As proven earlier through studies by dental morphometric measurements done by 2D image analysis can be performed by multiple operators with an excellent reliability.
4. Crown fabrication Wax-up for metal crowns was done with metal extension (25mm), to engage them in the Universal Testing Machine, using Dental Inlay casting wax (Inlay wax medium stick; GC-Dental Corp. Japan). The wax up was then invested using phosphate bonded gypsum material (GC-Super, Japan) and cast with Nickel-Chromium Ni-Cr metal alloy at the Prosthodontics laboratory of Fatima Jinnah Dental College. The cast crowns were then finished used metal finishing discs, making sure the metal extensions were not less than 20mm. The fitting surface of all crowns were sandblasted accordingly and were made ready for cementation process. The teeth were numbered between 1-120 for record purposes and random assignment to either of the study groups.
5. Cementation Tooth mounts were randomized using their serial numbers, to either of the three cement application techniques. This random allocation was done by generating a random sequence using Microsoft Excel by one of the department's lecturers, not directly related to the study. 40 teeth were allocated to each group. This sequence was passed on to an external operator (a general dentist), again not related to the primary research team, who was trained by the PI prior to study commencement on how to apply cement according to the operational definitions of the three cementation techniques under observation in this study. The cementation process started with mixing of permanent glass ionomer type-I luting cement (3M Ketac Cem Radiopaque Hand mix, USA) according to the manufacturer's recommendation by a single operator to ensure uniformity of mixing technique. The liquid component of Glass Ionomer Cement was measured using a 1cc syringe, while powder was measured using manufacturer provided scoop to ensure equal amount of cement was mixed. The mixing was done on a glossy paper pad provided by the manufacturer.

   The external operator cemented the metal crowns on the tooth mounts according to their allocation of cementation category. They were then seated by applying 80Newton pressure using a hydraulic press for 10 minutes. After ensuring the cement had dried completely the cemented crowns (on mounts) were left for seven days, soaked in distilled water to ensure hydration and to replicate intra-oral moisture conditions.
6. Testing for retention On the eighth day, the PI undertook the experiment of retention testing. To help in minimizing bias while performing the retention testing, the PI and field assistant did not know which cement application technique had been used under mounted tooth being observed. The two components (Tooth mount with cemented crown) were then attached to a Universal Testing Machine (INSTRON-4301) and tensile forces were applied to check the retention of the crown. The amount of force required was monitored on the computer. The force of traction was increased slowly till the crown de-bonded and came off the prepared tooth. That value of force in Newtons was noted in the proforma against the tooth mount's serial number. The entire procedure was done under supervision of a field assistant from Pakistan Council of Scientific and Industrial Research laboratory. PI was unblinded after completion of data analysis. The serial number allocation to study groups was directly conveyed to the statistician by the external observer. All data were recorded in pre-formed proforma.

ELIGIBILITY:
Inclusion Criteria:

* Second pre-molar tooth.
* Mandibular arch.
* Visibly sound tooth; without any pathology e.g. dental caries
* Extraction referred by Orthodontics Department.

Exclusion Criteria:

* Carious teeth.
* Fractured or broken teeth.
* Teeth with patient history of dental anomaly.
* Teeth with any restoration e.g. filling.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Cementation technique A,B and C | 9 months
  1. Filling the crown with cement up to margins.
  2. Applying a cement layer on all fitting surfaces.
  3. Applying a cement layer on all fitting surfaces except occlusal surface.
  Each of the aforementioned groups exhibits distinct measures of tensile strength. Each group will be compared with one another in terms of the cementation technique used, specifically in relation to Newton force.
  A questionnaire was not employed for comparative purposes among the three groups; instead, the unit of force (Newton) was utilized to compare each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Jinnah Dental College, Karachi, Sindh, Pakistan